CLINICAL TRIAL: NCT02802059
Title: E. Coli Nissle 1917 - Suspension for Infection Prophylaxis
Acronym: RONi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardeypharm GmbH (Industry)
Collaborators: ICON plc (Industry); Clinscience Sp. z o.o. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MU 1441; 2015-001763-39 (EudraCT Number)
Record Dates: First submitted 2016-01-18; First posted 2016-06-16 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-09

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EcN-Suspension (Experimental): 279 healthy functionally mature newborn infants up to 35 weeks gestational age, treated with EcN-Suspension
  Interventions: Drug: EcN-Suspension
- Placebo (Placebo Comparator): 279 healthy functionally mature newborn infants up to 35 weeks gestational age, treated with Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EcN-Suspension — Initial administration not later than 120h after birth. 14 ampoules a 1 ml are administered within a time of 3 weeks (1 ampoule per day within first week and 1 ampoule every second day within the following two weeks).
  Subsequent re-administration after 6 and 12 months. 10 ampoules a 1 ml are administered within 10 days (1 ampoule per day).
  Other Names: E. coli strain Nissle 1917 bacteria
  Arms: EcN-Suspension
Drug: Placebo — Initial administration not later than 120h after birth. 14 ampoules a 1 ml are administered within a time of 3 weeks (1 ampoule per day within first week and 1 ampoule every second day within the following two weeks).
  Subsequent re-administration after 6 and 12 months. 10 ampoules a 1 ml are administered within 10 days (1 ampoule per day).
  Arms: Placebo

SUMMARY:
This study evaluates the long term effects of E. coli strain Nissle 1917 (EcN-Suspension) probiotic bacteria administration on the number of both, bacterial and viral infections during the first 24 months of infant's life. Half of study participants will receive EcN-Suspension, while the other half will receive placebo. In an additional non-clinical explorative evaluation will furthermore be investigated whether the early intestinal colonization with E.coli strain Nissle 1917 affects the establishment of the intestinal microbiota.

DETAILED DESCRIPTION:
In the course of the present trial the participants will be observed during the first 24 months of life, starting right after birth.

All newborns meeting all inclusion criteria and non-fulfilling any exclusion criteria will be included into the trial. Each participant of this clinical trial will be randomly allocated to one of the two trial arms, by using the method of randomly permuted blocks.

The newborns will be primarily treated during the first three weeks of life and re-treated after 6 and 12 months according to trial interventional plan.

Data on the efficacy and safety will be recorded during control visits after first month, 6, 12, 18 and 24 months.

A follow-up examination of study participants will be performed two years after the end of the participation in the present trial (i.e. at an age of 48 months), during which each child will be examined for its normal physical and cognitive development (covered by the U8 standardized examination). In addition data on allergic/atopic complaints or symptoms will be recorded.

In an additional non-clinical explorative evaluation, it will furthermore be investigated whether the early intestinal colonization with E.coli strain Nissle 1917 affects the establishment of the intestinal microbiota. Therefore stool samples of study participants will be collected at an age of 24 and 48 months. The microbial composition of these samples will be characterized and compared between the two trial arms (EcN vs. placebo).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form by the parents
* Age at inclusion: max. 120 hours after birth
* Functionally mature infant
* Gestational age more than 35th week of development
* Mother's intention to breastfeed the participant
* Readiness of the mother to administer no probiotics additionally to the trial medication

Exclusion Criteria:

* Non-fulfilment of the at least one inclusion criteria
* Lack of propensity/compliance of mother
* 5 min APGAR SCORE less than 5
* 10 min APGAR SCORE less than 8
* pH of umbilical cord blood less than 7 (Determination not obligatory, if APGAR SCORES do not indicate that the child may have suffered from a perinatal asphyxia)
* Any perinatal infection required antibiotic treatment
* Birth weight less than 2000 g
* TORCH-infection of the mother
* HIV-infection of the mother
* Any severe medical condition of mother or newborn which in the opinion of the investigator may have a critical impact on the conduct of the study.

Max Age: 120 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 567 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Number of infections | during the first 24 months of life
  The total number of infections observed for each participant during its individual study participation standardised per month during the first 24 months of life.
  An infection is an episode of illness caused by:
  * Acute upper respiratory tract infections
  * Acute lower respiratory tract infections
  * Otitis media
  * Gastroenteritis
  * Urinary tract infections
  The duration of an episode of illness is defined as the time from the appearance of the first symptom of a study relevant infection to the disappearance of the last symptom. Infections that occur concurrently or one after another within a period of 7 days are only counted separately, if they belong to different groups of illness.
  All rhinitides that occur in the first year of a child's life are considered for the count of the primary efficacy variable. Rhinitides that occur in the second year will only be included if they were accompanied by fever (body temperature higher than 38.4°C during at least one measure).

SECONDARY OUTCOMES:
Severity of the course of infections considered as primary variables quantified as the "duration of infections" | during the first 24 months of infants' life
  duration of infection = the number of days with at least one symptom
Severity of the course of infections considered as primary variables quantified as the "number of hospital admissions caused by infections" | during the first 24 months of infants' life
  number of hospital admissions caused by infections
Severity of the course of infections considered as primary variables quantified as the "mean number of in-hospital spent days due to infections" | during the first 24 months of infants' life
  mean number of in-hospital spent days due to infections
Severity of the course of infections considered as primary variables quantified as the "number of antibiotic treatments due to infections". | during the first 24 months of infants' life
  number of antibiotic treatments due to infections
Severity of the course of infections considered as primary variables quantified as the "number of adverse events". | during the first 24 months of infants' life
  number of adverse events
Severity of the course of infections considered as primary variables quantified as the "tolerance to trial medication". | during the first 24 months of infants' life
  Tolerance of trial medication will be assessed by the investigator and scored "very good", "good", "moderate", or "poor".

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Wolff, Dipl-Biophys, Study Director — Ardeypharm GmbH; Dirk M Olbertz, MD, Principal Investigator — Klinikum Südstadt Rostock - Abteilung für Neonatologie
Locations (6):
- Germany (4):
  - Krankenhaus St. Elisabeth & St. Barbara, Halle
  - Universitätsklinikum Jena - Klinik für Kinder- und Jugendmedizin, Jena
  - Klinikum Westbrandenburg, Potsdam
  - Klinikum Südstadt Rostock - Abteilung für Neonatologie, Rostock
- Poland (2):
  - Oddział Kliniczny Noworodków, Wcześniaków z Intensywną Terapią Noworodka wraz z Wyjazdowym Zespołem "N", Bydgoszcz
  - Samodzielny Publiczny Dziecięcy Szpital Kliniczny Oddział Kliniczny Neonatologiiul, Warsaw

IPD SHARING:
Plan to Share IPD: No